CLINICAL TRIAL: NCT00615134
Title: A Randomized, Open-label Study Evaluating the Antiviral Activity and Safety of 3 Month Fuzeon Induction With an Optimized Background Antiretroviral Regimen Versus OB Alone, in Fuzeon-naive HIV-1 Infected Patients With Virological Failure.
Brief Title: INNOVE Study: A Study of 3 Months Induction With Fuzeon (Enfuvirtide) + Optimized Background (OB) Versus OB Alone in HIV-1 Infected Patients With Virological Failure.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21287
Record Dates: First submitted 2008-01-30; First posted 2008-02-14 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: HIV Infections
Keywords: treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: enfuvirtide [Fuzeon]; Drug: Optimized background ARV therapy
- 2 (Active Comparator)
  Interventions: Drug: Optimized background ARV therapy

INTERVENTIONS:
Drug: enfuvirtide [Fuzeon] — 90mg sc bid
  Arms: 1
Drug: Optimized background ARV therapy — As prescribed

SUMMARY:
This 2 arm study will assess the efficacy and safety of a new regimen of Fuzeon

+ optimized background antiretroviral treatment, in Fuzeon-naive HIV-1 infected patients with virological failure. Eligible patients will be randomized to recei ve either new optimized treatment alone, or optimized treatment + Fuzeon 90mg s.

c. twice daily, to determine the effect of 3 month induction with Fuzeon.It will be possible for a patient to receive several additional 3 month periods with F uzeon, in the case of new virological failure. The anticipated time on study tre atment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* HIV-1 infection, with virologic failure;
* on same stable HAART for >4 weeks, with viral load >1000 RNA copies/mL;
* Fuzeon-naive.

Exclusion Criteria:

* coinfection with HIV-2;
* active opportunistic infection in 4 weeks prior to screening;
* cirrhosis or severe liver failure;
* severe renal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with plasma viral load <50 copies/mL | Week 24

SECONDARY OUTCOMES:
CD4 count, virological responders, time to virological failure, number of Fuzeon 'sequences'/patient, AEs, ADEs, injection site reactions. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- France (26):
  - Aulnay-sous-Bois
  - Basse-terre
  - Bordeaux
  - Boulogne
  - Caen
  - Colmar
  - Fort-de-france
  - Garches
  - La Roche-sur-Yon
  - Le Kremlin-Bicêtre
  - Levallois-Perret
  - Lyon
  - Marseille
  - Nantes
  - Nice
  - Nîmes
  - Paris
  - Pessac
  - Pointe à Pitre
  - Poitiers
  - Pontoise
  - Rouen
  - Saint-Denis
  - Saint-Pierre
  - Toulouse
  - Tourcoing